CLINICAL TRIAL: NCT02674321
Title: A Pilot Study Of SD-809 (Deutetrabenazine) In Moderate To Severe Tourette Syndrome
Brief Title: A Pilot Study Of SD-809 (Deutetrabenazine) In Moderate To Severe Tourette Syndrome (TS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Auspex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SD-809-C-17
Record Dates: First submitted 2016-02-02; First posted 2016-02-04 (Estimated); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: TOURETTE SYNDROME
Keywords: Tourette Syndrome; adolescents
MeSH Terms: conditions — Tourette Syndrome | interventions — deutetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SD-809 (Experimental): • SD-809 tablets taken once or twice daily for 8 weeks, includes a dose titration period and a maintenance period.
  Interventions: Drug: SD-809

INTERVENTIONS:
Drug: SD-809

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and preliminary efficacy of SD-809 in the treatment of motor and phonic tics of Tourette Syndrome and to evaluate the pharmacokinetic of SD-809 and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18 years of age, inclusive, at Screening.
* Patient has a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) diagnosis of Tourette Syndrome and has manifested motor and phonic tics within 3 months before the Screening visit
* Patient has total tic score of ≥19 on the YGTSS
* Tic severity and frequency has been stable for at least 2 weeks before the Screening visit
* Willing to adhere to medication regimen and to comply with all procedures
* Patient is in good general health, as indicated by medical and psychiatric history and physical examination
* Patient and parent/guardian have provided written, informed consent (and written assent, as appropriate)
* Female patients of childbearing potential agree to use an acceptable method of contraception

  * Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* Patient has a serious untreated or undertreated psychiatric illness
* Patient has a history of suicidal ideation or behavior
* Patient has received tetrabenazine, neuroleptics, benzodiazepines, topiramate, dopamine receptor antagonists within 14 days of Screening or Baseline; or botulinum toxin within 3 months of Screening or Baseline
* Patient is being treated with deep brain stimulation for control of tics
* Patient has a progressive or degenerative neurological disorder or a structural disorder of the brain
* Patient has participated in an investigational drug or device trial within 30 days of Screening
* Patient is pregnant or breastfeeding at Screening or Baseline
* Patient has a history of alcohol or substance abuse in the previous 12 months, as defined in the DSM-V

  * Additional criteria apply, please contact the investigator for more information

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety | 8 weeks
  Incidence of adverse events (AEs), serious AEs, severe AEs, drug related AEs, AEs leading to withdrawal.

SECONDARY OUTCOMES:
Change from Baseline in Total Tic Score of the Yale Global Tic Severity Scale (YGTSS) | Baseline, Weeks 2, 4 and 8
Change from Baseline in Impairment Score of the Yale Global Tic Severity Scale (YGTSS) | Baseline, Weeks 2, 4, and 8
Change from Baseline in Global Severity Score of the Yale Global Tic Severity Scale (YGTSS) | Baseline, Weeks 2, 4, and 8
Change from Baseline in Tourette Syndrome Clinical Global Impression | Baseline, Weeks 2, 4, and 8
Patient Global Impression of Change (TS-PGIC) | Weeks 2, 4, and 8

OTHER OUTCOMES:
Pharmacokinetic parameters | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (1):
- Teva Investigational Site #101, Houston, Texas, United States